CLINICAL TRIAL: NCT00352196
Title: A Biological Basis of Therapy for Negative Symptom Spectrum Disorders: Risperdal Effect on Frontal Metabolism in Asperger's Disorder
Brief Title: Janssen Asperger's MRS (Magnetic Resonance Spectroscopy Risperidone Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Donna Londino, Associate Professor, Augusta University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIS-EMR-4026; MCG HAC File #01-09-063 (Other: Institutional Review Board)
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Asperger's Disorder
Keywords: Asperger's Disorder; Risperidone; Magnetic Resonance Spectroscopy; Social Skills
MeSH Terms: conditions — Asperger Syndrome; Social Skills | interventions — Risperidone; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnetic Resonance Spectroscopy (Experimental): Subjects will receive a baseline MRS prior to and within 7 day of completing 12 weeks of standard treatment with.
  Interventions: Drug: Risperidone; Other: Magnetic Resonance Spectroscopy
- NO-MRS (Other): Subjects will receive 12 weeks of standard treatment of risperidone 0.25 to 11 mg per day, or early termination. Dose titration will based on response and tolerability.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — 12 weeks of treatment with risperidone 0.25 to 11 mg per day.
  Other Names: Risperdal
Other: Magnetic Resonance Spectroscopy — Subjects will receive a standard MRS to assess the concentrations and ratios of brain metabolites N-acetylaspartate, creatine, phosphocreatine, and choline.
  Other Names: MRS
  Arms: Magnetic Resonance Spectroscopy

SUMMARY:
This study will be an open-label, 12-week trial of risperidone in subjects with Asperger's Disorder, according to Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) Criteria. The study has two arms, one involving pre- and post-treatment MRS studies, and one without MRS. The MRS arm will study 18-20 subjects ages 6 and above, with a target of 14 completing patients. For both arms, we plan to a enroll at total of 30 patients to achieve completion for 24 patients. The non-MRS arm of the study will include subjects 6-18 years of age, the bulk of which have completed the study as of the writing of this updated revision. Our hypotheses are that treatment of Asperger's patients with a low dose of risperidone will:

1. decrease ratios of N-acetylaspartate (NAA), creatine, phosphocreatine (Cr + PCr), and choline in the prefrontal lobe, and
2. decrease the severity of negative symptoms and overall improve social behavior, and
3. that the two will be correlated.

Specific Aims

The primary objectives of this trial are to:

* Further assess and investigate the utility of risperidone in the treatment Asperger's disorder.
* Assess the efficacy of risperidone in normalizing increased frontal lobe metabolites.
* Assess the efficacy of risperidone in normalizing symptoms in Asperger's disorder patients using standardized rating scales to assess the impact on negative symptoms and on social interaction.
* Determine whether risperidone's effect on clinical improvement of Asperger's disorder, i.e., negative symptoms, is correlated with normalization of frontal lobe metabolites
* Accrue safety and tolerability data on risperidone for this population of patients.

This information could potentially be used to provide pilot data for a double blind trial

DETAILED DESCRIPTION:
STUDY DESIGN

This study will be an open-label, 12-week trial of risperidone in subjects with Asperger's Disorder, according to DSM-IV Criteria. The study has two arms, one involving pre- and post-treatment MRS studies, and one without MRS. The MRS arm will study 18-20 subjects ages 6 and above, with a target of 14 completing patients. For both arms, we plan to a enroll at total of 30 patients to achieve completion for 24 patients. The non-MRS arm of the study will include subjects 6-18 years of age, the bulk of which have completed the study as of the writing of this updated revision.

Subjects will first undergo a screening visit during which safety and diagnostic assessments are completed, and a minimum of 3 days will be allowed to evaluate the screening results. Then, the subjects will complete one or two practice sessions to provide training to achieve the necessary stillness for a duration that is sufficient to complete a MRS session. Upon completion of successful practice sessions, subjects will then be scheduled for a MRS visit. Once the MRS is successfully completed, subjects will be assigned to receive risperidone 0.25 mg at their baseline visit.

Response to risperidone will be measured at weeks 3, 6, 9, and 12 by the Scale for Assessment of Negative Symptoms (SANS). Additional secondary outcome measures are shown below (figure 1). A post-treatment MRS will be conducted after the Week 12 or early termination visit. Subjects will be given adequate medication supply to cover through the day of the final MRS visit.

Study Medication. Because Asperger's Disorder is diagnosed in childhood and is considered a childhood disease, our previous phase of the study focused on subjects ages 6 - 18. Published dosages of risperidone used in child, adolescent, and adult studies ranges from 0.25 to 11 mg per day. Most studies in children and adolescents begin with a starting dose of 0.25 mg bid, which is also appropriate for adults, and will be the starting dose planned for this study. The study progresses from a fixed to a titrated dose paradigm. After Week 6, dose will be increased (based on response and tolerability), ranging from one to two tablets twice daily (either 1 or 2 mg of risperidone daily). Again at Week 9, dose will be increased (based on response and tolerability), ranging from 1 mg to 4 mg per day of risperidone, one to four tablets twice a day of risperidone. Patients who have any trouble tolerating the starting dose may have their dose reduced to 0.25 mg per day and continue in the study. Patients who cannot tolerate the 0.25 mg dosage would discontinue the study in order to receive alternative treatment.

Schedule of Events and Observations

Screening Visit: A Structured Clinical Interview for Diagnosis (SCID) in conjunction with DSM-IV criteria and a psychiatric history, will allow the study physicians to establish and confirm a diagnosis of Asperger's disorder. Medical history, vital signs, clinical labs {chemistry, complete blood count (CBC), thyroid function, urinalysis, urine drug screen, and blood pregnancy test (fecund females only)}, a physical exam, and an EKG will be performed to determine patient safety.

Blood Draws: Additional lab samples will be collected at both screening and end of study to explore 1) the effects of diet on treatment outcomes with risperidone, and 2) effects of risperidone treatment on levels of Brain Derived Neurotrophic Factor (BDNF) and Nerve Growth Factor (NGF). The additional blood will amount to an approximate total of 8 tablespoons of blood collected during the study.

MRS Visits and Practice Sessions: Subjects enrolling in the MRS arm, will be scheduled for a pretreatment MRS which will take place after the screening visit but before the baseline visit and prior to starting risperidone. Subjects will also have a post-treatment MRS within 7 days of their week 12 visit or at study termination. Patients will be supplied with enough medication to continue treatment until the MRS measures are complete.

Subjects may be required, based on the investigator's discretion, to complete one or two sessions during the screening period for Practice Sessions for MRS studies to better prepare subjects for the level of stillness needed for MRS studies. The practice sessions will last approximately one hour and will be performed at the Medical College of Georgia (MCG) Office of Clinical Investigative Services, located at 1521 Pope Ave, Suite FF-100. Practice Sessions may also be performed at the MRI suite at MCG to allow the subject to see or lie in the MRI machine, depending on availability.

Rationale for practice sessions: We have learned that these sessions may be necessary to help subjects achieve the stillness required for MRS. During the sessions, subjects will be trained to remain still while lying on a padded stretcher, using behavioral and relaxation training techniques performed by a qualified investigator. Other efforts will be made to simulate the MRS environment that may include playing recorded sounds of a MRI machine and simulation of the padded head supports.

In most cases the Practice Sessions, would be all done prior to the MRS visit, but in some cases of a failed MRS visit, the investigator may choose to schedule another practice session prior to re-trying the MRS visit. The practice session will supplement the standard efforts used to support patients' compliance during MRI procedures. For example, part of the hospital's usual care during MRI studies includes the option of having the patient wear video goggles and headphones. Subjects in our study may view a calming video of neutral content to aid in problems affecting stillness.

Behavioral reinforcement and subject payments during practice sessions. Part of the payment for practice sessions will be used as a behavioral reinforcement plan, and this will be in addition to the $20 payment for clinic visits, reimbursement for travel over 25 miles one-way @ .28/mile, and $50 for the MRS visit (paid regardless of success or failure).

The additional subject payment in the practice session will be used as incentive and behavioral reinforcement for achieving stillness. Specifically, subjects will receive a token (such as a poker chip or printed paper token) worth $5.00 for each 5-minute period they remain still. If a subject's head moves during a period, they will be told they have to begin a new period. The achievement of stillness will be determined by the investigator at the time, taking into account the actual observed stillness and the need to encourage and reward the subjects' efforts.

The actual stillness practice will last up to 40 minutes, and the subject will receive a token for each 5 minute period they remain still, for up to 8 periods. The total additional payment for behavioral reinforcement will range from $5.00 to $40.00, to be paid in the same way as other subject payments. In the case of adolescent subjects, parents will be encouraged to consider the additional practice session payments to go to the child as a reward for the child's efforts.

Baseline Visit: Subjects will be scheduled for baseline procedures when lab results and MRS values are reviewed and approved by the study physician, in most cases expected to be a period of 7 days. This visit will consist of medical-psychiatric interviews and neurocognitive testing. A urine pregnancy test (done previously at screening) may be repeated at baseline based on the judgement of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be age 6 -18 for the Non-MRS arm of the study, and age 6 or above for the MRS arm of the study.
2. If applicable, a parent or legal guardian or legal representatives of study subject must provide informed consent and sign an informed consent document.
3. Female patients of childbearing age must be either postmenopausal for at least one year, surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (oral or parenteral hormonal contraceptives, intrauterine device; barrier and spermicide. Abstinence is not an acceptable method).
4. Female patients of child-bearing potential must have a negative pregnancy test to be performed at screening and baseline.
5. Patients must meet DSM-IV criteria for Asperger's Disorder. Other Axis I & II disorders excluded are listed below.
6. Patient must not have other serious, unstable illnesses and must be otherwise physically healthy on the basis of a physical examination, medical history, electrocardiogram and the results of blood biochemistry, hematology tests and a urinalysis.
7. Patient must have a negative urine drug screen with the exception of amphetamines if the patient is being treated with stimulants for four months or longer prior to entry.

Exclusion Criteria:

1. Patients who meet DSM-IV criteria for any psychotic disorder including schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, shared psychotic disorder, psychotic disorder due to a general medical condition, substance-induced psychotic disorder,psychotic disorder not otherwise specified, major depression with psychotic features, or bipolar disorder.
2. Patients who meet DSM-IV criteria for schizoid, schizotypal, or paranoid personality disorder. Patients who meet DSM-IV criteria for autistic disorder or pervasive developmental disorder.
3. Claustrophobic patients and those otherwise unable to successfully complete the MRS procedure prior to baseline.
4. Patients who meet criteria for substance abuse or dependence within the past three months. (Nicotine and caffeine are exceptions).
5. Patients believed by the investigator to be at significant risk for suicidal or violent behavior during the course of the trial.
6. Female patients who are pregnant or nursing.
7. Patients with a known or suspected seizure disorder.
8. If the results of the serum alanine transaminase (ALT) or aspartate aminotransferase (AST) are more than twice the upper limit of the central laboratory's reference range, the patient may not be enrolled. If the results of any other biochemistry, hematology or urinalysis tests are not within the central laboratory's reference ranges, the patient can be enrolled only on condition that the investigator judges that the deviations are not clinically significant. This should be clearly recorded on the laboratory report and in the source documents.
9. Patients with a history of neuroleptic malignant syndrome (NMS) or similar encephalopathic syndrome.
10. Patients who, by history, have received treatment with Risperdal or another neuroleptic (including olanzapine or quetiapine) within three months of baseline evaluation. Patients who have received a depot antipsychotic within one treatment cycle prior to screening. Patients who have taken an antidepressant, or lithium within 4 weeks of the trial, 6 weeks for fluoxetine. Patients who have taken any psychotropic medication within 1 week of the trial. Patients who require concomitant medications during the trial.
11. Patients with a suspected history of hypersensitivity or intolerance to risperidone.
12. Patients with a known or suspected history of severe drug allergy or hypersensitivity (e.g., Steven Johnson's syndrome)
13. Patients with an anticipated life expectancy of six months or less.

    -

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Chang in the Scale for the Assessment of Negative Symptoms (SANS) | Baseline, Week 3, 6, 9, 12 and up to 7 weeks post treatment

SECONDARY OUTCOMES:
Change in Positive and Negative Symptom Scale (PANNS) | Baseline, Week 3, 6, 9, 12 and up to 7 weeks post treatment
Change in Brief Psychiatric Rating Scale (BPRS) | Baseline, Week 3, 6, 9, 12 and up to 7 weeks post treatment
Change in Montgomery Asberg Rating Scale (MADRS) | Baseline, Week 3, 6, 9, 12 and up to 7 weeks post treatment
Change in Global Assessment Scale (GAS) | Baseline, Week 3, 6, 9, 12 and up to 7 weeks post treatment
Change in Abnormal Involuntary Movement Scale (AIMS) | Baseline, Week 3, 6, 9, 12 and up to 7 weeks post treatment
Change in Neurocognitive test battery | Baseline, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Rausch, MD, Principal Investigator — Augusta University; Donna L Londino, MD, Study Director — Augusta University
Locations (1):
- Medical College of Georgia, Dept. of Psychiatry, Augusta, Georgia, United States